CLINICAL TRIAL: NCT00892814
Title: Partial Breast Versus Whole Breast Irradiation to Women ≥ 60 Years Operated With Breast Conservation for Early Breast Cancer: a Randomized Fase II Trial
Brief Title: Partial Breast Versus Whole Breast Irradiation in Elderly Women Operated on for Early Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Birgitte Offersen, M.D., Ph.D., ass. professor, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG PBI protocol; CIRRO IP030109
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Partial breast irradiation (Experimental): 40 Gy/15 fractions, 3 weeks
  Interventions: Radiation: Partial breast irradiation
- Whole breast irradiation (Active Comparator): 40 Gy/15 fractions, 3 weeks
  Interventions: Radiation: Whole breast irradiation

INTERVENTIONS:
Radiation: Partial breast irradiation — 40 Gy/15 fractions, 3 weeks
  Arms: Partial breast irradiation
Radiation: Whole breast irradiation — 40 Gy/15 fractions, 3 weeks
  Arms: Whole breast irradiation

SUMMARY:
The purpose of this trial is to investigate the difference in late radiation morbidity between partial breast irradiation and whole breast irradiation given to women operated on with breast conservation surgery for early breast cancer with a low risk of local recurrence.

DETAILED DESCRIPTION:
The study is 2-armed. In both treatment arms the radiotherapy consists of 40 Gy in 15 fractions, 2.67 Gy per fraction. The primary endpoint in the trial is late radiation morbidity evaluated as fibrosis, secondary endpoints are other types of late morbidity, rate of local recurrence and an attempt to establish a genetic risk profile for development of late radiation morbidity.

The hypothesis is that women operated with breast conservation for a breast carcinoma with low risk of local recurrence can be offered partial breast irradiation without risking more late radiation morbidity compared to whole breast irradiation.

ELIGIBILITY:
Inclusion Criteria:

* women 60 years or older
* operated for unilateral, unifocal early breast cancer pT1, pN0, M0, grade I or II, positive estrogen and/or progesterone receptor, HER2 negative

Exclusion Criteria:

* lobular carcinoma

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2009-05-14; Primary Completion 2016-03-07 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Grade 2 and/or 3 fibrosis after radiotherapy | 3 years

SECONDARY OUTCOMES:
Any other late morbidity after adjuvant radiotherapy, genetic risk profile for late morbidity, recurrence/survival | 10 years
  morbidity and recurrences

CONTACTS AND LOCATIONS:
Overall Officials: Lars Stenbygaard, MD, Study Chair — Aalborg University Hospital; Erik Jacobsen, MD, Study Chair — Vejle Hospital; Mette H Nielsen, MD, phd, Study Chair — Odense University Hospital; Anders N Pedersen, MD, phd, Study Chair — Rigshospitalet, Denmark; Birgitte Offersen, MD, phd, Principal Investigator — Aarhus University Hospital
Locations (1):
- The Danish Breast Cancer Cooperative Group, Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- [Background] Offersen BV, Overgaard M, Kroman N, Overgaard J. Accelerated partial breast irradiation as part of breast conserving therapy of early breast carcinoma: a systematic review. Radiother Oncol. 2009 Jan;90(1):1-13. doi: 10.1016/j.radonc.2008.08.005. Epub 2008 Sep 8. PMID 18783840
- [Derived] Offersen BV, Alsner J, Nielsen HM, Jakobsen EH, Nielsen MH, Stenbygaard L, Pedersen AN, Thomsen MS, Yates E, Berg M, Lorenzen EL, Jensen I, Josipovic M, Jensen MB, Overgaard J; Danish Breast Cancer Group Radiotherapy Committee. Partial Breast Irradiation Versus Whole Breast Irradiation for Early Breast Cancer Patients in a Randomized Phase III Trial: The Danish Breast Cancer Group Partial Breast Irradiation Trial. J Clin Oncol. 2022 Dec 20;40(36):4189-4197. doi: 10.1200/JCO.22.00451. Epub 2022 Aug 5. PMID 35930754